CLINICAL TRIAL: NCT05573477
Title: A Randomized, Active-controlled, Double-blind, Parallel, Multi Center, Phase 3 Study to Evaluate the Efficacy and Safety of Co-administrated ATB-1011 and ATB-1012 in Patients With Essential Hypertension and Type II Diabetes Mellitus
Brief Title: Evaluation of Efficacy and Safety of ATB-1011+ATB-1012 Co-administration for Essential Hypertension and Type II Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Autotelicbio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATB-101-003
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Essential Hypertension; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Essential Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1:1:1 ratio to 4 treatment arms. After completion of treatment period, participants will enter 12-week extension period and take 1 tab/day of ATB-1011 and ATB-1012.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ATB-1011 + ATB-1012 (Experimental): Participants will receive 1 tablet/day of each drug for 12 weeks
  Interventions: Drug: ATB-1011; Drug: ATB-1012; Drug: ATB-1013 placebo
- ATB-1012 + ATB-1013 (Experimental): Participants will receive 1 tablet/day of each drug for 12 weeks
  Interventions: Drug: ATB-1012; Drug: ATB-1013; Drug: ATB-1011 placebo
- ATB-1011 (Active Comparator): Participants will receive 1 tablet/day of each drug for 12 weeks
  Interventions: Drug: ATB-1011; Drug: ATB-1012 placebo; Drug: ATB-1013 placebo
- ATB-1012 (Active Comparator): Participants will receive 1 tablet/day of each drug for 12 weeks
  Interventions: Drug: ATB-1012; Drug: ATB-1011 placebo; Drug: ATB-1013 placebo

INTERVENTIONS:
Drug: ATB-1011 — Oral tablet
  Arms: ATB-1011; ATB-1011 + ATB-1012
Drug: ATB-1012 — Oral tablet
  Arms: ATB-1011 + ATB-1012; ATB-1012; ATB-1012 + ATB-1013
Drug: ATB-1013 — Oral tablet
  Arms: ATB-1012 + ATB-1013
Drug: ATB-1011 placebo — Placebo matched to ATB-1011
  Arms: ATB-1012; ATB-1012 + ATB-1013
Drug: ATB-1012 placebo — Placebo matched to ATB-1012
  Arms: ATB-1011
Drug: ATB-1013 placebo — Placebo matched to ATB-1013
  Arms: ATB-1011; ATB-1011 + ATB-1012; ATB-1012

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of ATB-1011 and ATB-1012 co-administration in patients with essential hypertension and type II diabetes mellitus

DETAILED DESCRIPTION:
Primary Objectives:

* To demonstrate superiority of 12-week co-administration of ATB-1011 and ATB-1012 in blood pressure control over ATB-1012 monotherapy
* To demonstrate superiority of 12-week co-administration of ATB-1011 and ATB-1012 in diabetes control over ATB-1011 monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Those with Primary Hypertension and Type II Diabetes Mellitus (DM)
* Those who have been given adequate explanation about the purpose and the details of the clinical trial and have given voluntary, written informed consent
* Those who have not taken any antihypertensive agents for ≥2 weeks prior to randomization.
* Those who have not taken any oral hypoglycemic agents, except for same dose of metformin (≥1000 mg/day), for ≥8 weeks prior to randomization

Exclusion Criteria:

* Those with reference arm mean sitting diastolic blood pressure (MSDBP) ≥110 mmHg at screening or at randomization
* Those with differences of systolic blood pressure (SBP) ≥ 20 mmHg and diastolic blood pressure (DBP) ≥ 10 mmHg between arms measured 3 consecutive times with ≥2 minutes between each measurement at screening
* Those with a history of alcohol or substance abuse
* Those who are pregnant or nursing
* Those who have received other clinical trial drugs within 12 weeks prior to screening
* Those who are deemed ineligible to participate in the clinical trial based on the medical opinion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Mean sitting systolic blood pressure (MSSBP) (ATB-1011+ATB-1012 vs. ATB-1012) | baseline to Week 12
  Change in MSSBP with ATB-1011 + ATB-1012 co-administration compared to ATB-1012 monotherapy
Hemoglobin A1c (HbA1c) (ATB-1011+ATB-1012 vs. ATB-1011) | baseline to Week 12
  Changes in HbA1c with ATB-1011 + ATB-1012 co-administration compared to ATB-1011 monotherapy

SECONDARY OUTCOMES:
MSSBP (ATB-1011+ATB-1012 vs. ATB-1011) | baseline to Week 12
  Changes in MSSBP with ATB-1011 + ATB-1012 co-administration compared to ATB-1011 monotherapy
MSSBP (ATB-1012+ATB-1013 vs. ATB-1012) | baseline to Week 12
  Changes in MSSBP with ATB-1012 + ATB-1013 co-administration compared to ATB-1012 monotherapy
MSSBP (ATB-1012+ATB-1013 vs ATB-1011+ATB-1012) | baseline to Week 12
  Changes in MSSBP with ATB-1012 + ATB-1013 co-administration compared to ATB-1011 + ATB-1012 co-administration
HbA1c (ATB-1011+ATB-1012 vs. ATB-1012) | baseline to Week 12
  Changes in HbA1c with ATB-1011 + ATB-1012 co-administration compared to ATB-1012 monotherapy
Changes in MSSBP | baseline to Weeks 4 and 8
Changes in mean sitting diastolic blood pressure (MSDBP) | baseline to Weeks 4, 8, and 12
Changes in HbA1c | baseline to Weeks 4, 8, and 12
Changes in glycemic parameters | baseline to Weeks 4, 8, and 12
  Fasting plasma glucose (FPG)
Changes in glycemic parameters | baseline to Weeks 4, 8, and 12
  Homeostatic model assessment of beta cell function (HOMA-beta)
Changes in glycemic parameters | baseline to Weeks 4, 8, and 12
  Homeostatic model assessment of insulin resistance (HOMA-IR)

OTHER OUTCOMES:
Extension period: Changes in HbA1c | baseline and Week 12 to Weeks 18 and 24
Extension period: Changes in MSSBP | baseline and Week 12 to Weeks 18 and 24
Extension period: Changes in MSDBP | baseline and Week 12 to Weeks 18 and 24

CONTACTS AND LOCATIONS:
Overall Officials: James Jun, MD, Study Director — Autotelicbio
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No